

# Fondazione Italiana Linfomi ONLUS

Sede legale: piazza Turati 5, 15121 – Alessandria
P.IVA IT 02143940068 C.F. 96039680069
Uffici Studi FIL: c/o Uffici PACTO, Spalto Marengo 44, 15121, Alessandria
Tel. 0131– 033153, Fax 0131 - 263455; e-mail: startup@filinf.it; sito web: www.filinf.it

Study ID: FIL GAEL

**Eudract Number: 2014-005697-10** 

ClinicalTrials.gov Identifier: NCT02495454

**Title:** GA101-miniCHOP regimen for the treatment of elderly unfit patients with diffuse large B-cell non-Hodgkin's lymphoma. A phase II study of the Fondazione Italiana Linfomi (FIL).

Final Study Report: version 1, April 30<sup>th</sup>, 2020



# FINAL STUDY REPORT

| Name of | Fondazione Italiana Linfomi ONLUS (FIL) |
|---|---|
| Sponsor/Company: | |
| S4 1 4 | |
| Study type: | Interventional/clinical study |
| Study phase: | II |
| Study title: | GA101-miniCHOP regimen for the treatment of elderly unfit patients with |
| | diffuse large B-cell non-Hodgkin's lymphoma. A phase II study of the |
| | Fondazione Italiana Linfomi (FIL). |
| EudraCT: | 2014-005697-10 |
| ID study: | FIL_GAEL |
| Version: | 1 |
| Date: | September 29 <sup>th</sup> , 2014 |
| Name of Active | |
| Ingredient: | Cyclophosphamide |
| | Doxorubicin |
| | Vincristine |
| | Prednisone |
| <b>Conditions (diagnosis):</b> | Elderly unfit patients with CD20 positive Diffuse Large B-cell Lymphoma and |
| , 3 | Follicular grade IIIB, according to WHO classification |
| Studied period (years): | |
| CA authorization: | 24/04/2015 |
| lead EC opinion date: | 25/03/2015 |
| date of first enrolment: | 25/08/2015 |
| date of last completed: | 19/02/2020 |
| date of Interim Analysis | 22/03/2017 |
| (If applicable): | 22/03/2017 |
| (ii upplicuote). | |
| Study coordinator: | |
| | Francesco Merli, MD: |
| | Azienda Unita Sanitaria Locale-IRCCS - Arcispedale Santa Maria Nuova |
| | Ematologia – Reggio Emilia |
| Study centres: | |
| | Manuela Zanni, MD: |
| | A.O. SS. Antonio e Biagio e Cesare Arrigo - S.C. Ematologia - Alessandria |
| | Guido Gini, MD: |
| | AOU Ospedali Riuniti - Clinica di Ematologia - Ancona |
| | Annarita Conconi, MD |
| | Ospedale Degli Infermi - S.C. Oncologia - Biella |
| | Alessandra Tucci, MD |
| | ASST Spedali Civili di Brescia – Ematologia - Brescia |
| | Gerardo Musuraca, MD |
| | Istituto Scientifico Romagnolo per lo Studio e la Cura dei Tumori (I.R.S.T.) – |
| | Ematologia - Meldola |



| | Paola Matteucci, MD |
|---|---|
| | Fondazione IRCCS Istituto Nazionale dei Tumori di Milano – Ematologia <b>Milano</b> |
| | Samantha Pozzi, MD |
| | Azienda Ospedaliero-Universitaria Policlinico di Modena - Dipartimento Scienze Mediche e Chirurgiche Materno-Infantili e dell'Adulto - <b>Modena</b> |
| | Gianluca Gaidano, Prof. |
| | AOU Maggiore della Carita di Novara - SCDU Ematologia - Novara |
| | Dario Marino, MD |
| | I.R.C.C.S. Istituto Oncologico Veneto - Oncologia 1 – Padova |
| | Maurizio Musso, MD |
| | Casa di Cura La Maddalena - Oncoematologia e TMO Dip. Oncologia - Palermo |
| | Claudia Cellini, MD |
| | Ospedale delle Croci – Ematologia - Ravenna |
| | Annalia Molinari, MD |
| | Ospedale degli Infermi di Rimini - U.O. di Ematologia - Rimini |
| | Anna Marina Liberati, Prof.ssa |
| | A.O. S. Maria di Terni - S.C. Oncoematologia - Terni |
| | Federica Cavallo, MD |
| | A.O.U. Città della Salute e della Scienza di Torino - Ematologia Universitaria - <b>Torino</b> |
| | Merli Michele, MD |
| | Ospedale di Circolo - U.O.C Ematologia - Varese |
| Date of last database download: | e 27/04/2020 |
| Report date: | 30/04/2020 |
| • | |
| | List of abbreviations |
| | ADL Activity of Daily Living |
| | AE Adverse Events |
| | ALC Absolute Lymphocyte Count |
| | ALT Alanine Aminotransferase |
| | ASC Aspartate Aminotransferase |
| | ASCO American Society of Clinical Oncology |
| | B2M Beta2-microglobuline |
| | BM Bone Marrow |
| | CGA Comprehensive Geriatric Assessment |
| | CHOP Cyclophosphamide, Doxorubicin, Vincristine, Prednisone |
| | CI Confidence interval |
| | CIRS Cumulative Illness Rating Scale |



| | CNIC | C + 1N C + |
|---|---|---|
| | CNS | Central Nervous System |
| | CR | Complete Remission |
| | CRR | Complete Remission Rate |
| | CT scan | Computed Tomography Scan |
| | CTCAE | Common Terminology Criteria for Adverse Events |
| | DLBCL | Diffuse Large B Cell Lymphoma |
| | ECOG | Eastern Cooperative Oncology Group |
| | EORTC | European Platform of Cancer Research |
| | FDG-PET | Fluorodeoxyglucose Positron Emission Tomography |
| | FIL | Fondazione Italiana Linfomi |
| | FU | Follow Up |
| | GA101 | Obinutuzumab |
| | G-CSF | Granulocyte Colony-Stimulating Factor |
| | Hb | Hemoglobin |
| | HBcAb | Hepatitis B Core Antibody |
| | HBsAg | Hepatitis B surface antigen |
| | HCV | Hepatitis C Virus |
| | HIV | Human Immunodeficiency Virus |
| | I | Initial |
| | IADL | Instrumental Activity of Daily Living |
| | ISRT | Involved Site Radiation Therapy |
| | IPI | International Prognostic Index |
| | LVEF | Left Ventricular Ejection Fraction |
| | MEDdra | Medical Dictionary for Regulatory Activities |
| | ORR | Overall Response Rate |
| | OS | Overall Survival |
| | PET | Positron Emission Tomography |
| | PFS | Progression Free Survival |
| | PR | Partial Remission |
| | PRR | Partial Response Rate |
| | QoL | Quality of Life |
| | SAE | Serious Adverse Event |
| | SD | Stable Disease |
| | SUSAR | Suspected Unexpected Serious Adverse Reaction |
| | TLBCL | T-cell/histiocyte LBCL |
| | ULN | Upper Limit of Normality |
| | WBC | White Blood Cell |
| | WHO | World Health Organization |
| Study description (Aim of the study) | | |
| Primary objectives | The primary ob | jective is to assess whether the regimen GA101-miniCHOF |
| , , | | plute increase of the CR proportion of at least 15% (from 60% |
| | | 6 respect to R-miniCHOP regimen. To evaluate the activity of GA101- |
| | | miniCHOP regimen in terms of complete response rate (CRR) |
| Secondary objectives: | | e safety and tolerability of GA101 miniCHOP regiment |
| , , | in terms of adver | |
| | - Partial and Ove | erall Response Rate: PR and ORR (CR+PR) |
| | - Overall Survival (OS) | |
| | - Progression Free Survival (PFS) | |



| | - Dynamics of Comprehensive Geriatric Assessment (CGA) |
|---|---|
| | - Dynamics of Quality of Life (QoL) questionnaires |
| Primary end-points: | Complete Response Rate after 10 infusions of GA101 and 6 cycles of miniCHOP. The response rate to therapy will be based a central Independent |
| | Review Committee of response that will not consider the results of FDG-PET |
| | but will only use the conventional CT scan images (International Criteria, B. |
| | Cheson, JCO 1999) |
| Secondary end-points: | - Rate of Adverse Events |
| | - Partial and Overall Response Rate (PRR, ORR) |
| | - Overall Survival (OS) |
| | - Progression Free Survival (PFS) |
| | - Change in ADL, IADL and CIRS |
| TIL 11 1114 14 1 | - Change in QoL (EORTC QLQ C30) |
| Eligibility criteria | 1) 11' 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 |
| Inclusion | 1) Histologically proven CD20 positive Diffuse Large B-cell Lymphomaan |
| | Follicular grade IIIB lymphoma, according to WHO classification (local |
| | pathologist) |
| | 2) Age $\geq$ 65 years |
| | 3) No previous treatment |
| | 4) CGA assessment performed before starting treatment |
| | 5) UNFIT patients defined as follows |
| | - Age > 80 years with FIT profile, i.e. |
| | - ADL =6 residual functions |
| | - IADL=8 residual functions |
| | - CIRS: no comorbidity of grade 3-4 and <5 of grade 2 or Age < 80 with UNFIT profile, i.e |
| | - ADL > 5 residual functions |
| | - IADL > 6 residual functions |
| | - CIRS: no comorbidity of grade 3-4 and 5-8 co-morbidities of grade 2 |
| | 6) Ann Arbor Stage I with bulky, II-IV |
| | 7) At least one bi-dimensionally measurable lesion defined as > 1.5 cm in its |
| | largest dimension on CT scan |
| | 8) ECOG performance status of 0, 1, or 2 |
| | 9) Adequate hematologic function (unless caused by bone marrow infiltrat defined as follows: |
| | - Hemoglobin ≥ 10 g/dL |
| | - Absolute neutrophil count $\geq 1.5 \times 10^9/L$ |
| | - Platelet count $\geq 100 \times 10^9/L$ |
| | 10) LVEF >50% |
| | 11) Ability and willingness to comply with the study protocol procedure |
| | 12) Life expectancy > 6 months |
| | 13) Accessibility of patient for treatment and follow up |
| | 14) Written informed consent |
| Exclusion | 1) History of severe allergic or anaphylactic reactions to humanized or murine |
| 2. Total of | monoclonal antibodies or known sensitivity or allergy to murine products |
| | 2) Contraindication to any of the individual components of CHOP, including |
| | prior receipt of anthracyclines |
| | 3) History of other malignancies within 5 years prior to study entry except for |
| | adequately treated carcinoma in situ of the cervix or basal or squamous cell skin |
| | cancer |
| | 4) Stage I without bulky |
| | 5) Patients with transformed lymphoma |



| | 6) Prior therapy for DLBCL, with the exception of nodal biopsy or local |
|---|---|
| | irradiation |
| | 7) Previous exposure to cytotoxic agents |
| | 8) Suspect or clinical evidence of CNS involvement by lymphoma |
| | 9) HBsAg, HCV or HIV positivity; isolated HBcAb positivity is accepted only |
| | with concomitant treatment with Lamivudine |
| | 10) AST /ALT > twice upper the normal range; bilirubin > twice upper the |
| | normal range; serum creatinine > 2.5 mg/dl (unless these abnormalities were |
| | related to the lymphoma) |
| | 11) Evidence of any severe active acute or chronic infection |
| | 12) Concurrent co-morbid medical condition which might exclude |
| | administration of full dose chemotherapy |
| Treatments description | |
| | 6 courses of GA101-miniCHOP regimen and 2 additional infusions of |
| | GA101, every 21 days (for a total of 6 courses of miniCHOP and 10 infusions |
| | of C(1101) |

of GA101)

## **GA101-miniCHOP** regimen

#### Cycle 1

GA101: 1000 mg day 1, day 8 and day 15, iv Cyclophosphamide: 400 mg/mq, day 1, iv

Doxorubicin: 25 mg/mq, day 1, iv Vincristine: 1 mg, day 1, iv Prednisone: 40 mg/mq, days 1-5, os

#### Cycles 2-6

GA101: 1000 mg day 1, iv

Cyclophosphamide: 400 mg/mq, day 1, iv

Doxorubicin: 25 mg/mq, day 1, iv Vincristine: 1 mg, day 1, iv Prednisone: 40 mg/mg, days 1-5, os

Two additional infusions of GA101: 1000 mg day 1, iv, every 21 days.

Prophylactic granulocyte colony-stimulating factor (G-CSF) support is mandatory starting within 24-72 hours from day 1 of each cycle for no less than 4 doses or until neutrophils count exceeds 1.00×10°/L or more (ASCO guidelines JCO - 2006). Alternatively, a single dose of pegylated G-CSF br pegfilgrastim can be used.

Use of erythropoietin is allowed according to clinical practice.

A preliminary debulking or symptomatic phase of vincristine 1 mg or intermediate -- high dose steroid is allowed.

In case of debulking with vincristine, this drug must be omitted from cycle1.

## Involved Site Radiotherapy (ISRT) is allowed on previous bulky sites or on PET positive lesion at the end of treatment.

An interim check for response will be assessed after the completion of 4 courses of GA101-miniCHOP in order to identify nonresponding patients: patients achieving a CR, PR, or SD will continue to complete combined immunochemotherapy as planned, patients with progressive disease will stop treatment and will be considered as failure.



All patients stopping study treatment due to early disease progression will be followed for survival until the end of the study.

#### Dosage Delays and Modifications: GA101 and CHOP chemotherapy

Dose reductions and delays are based on all laboratory values obtained within 72 hours prior to a study treatment infusion.

A dose delay of 21 days is permitted for miniCHOP and GA101 to allow recovery of hematologic toxicities to Grade  $\leq$  2 (platelets must return to Grade  $\leq$  1) or non-hematologic toxicities to Grade  $\leq$  1 or baseline status for the first episode.

### Dose Modifications of GA101-miniCHOP chemotherapy

No dose modifications of GA101 (1000 mg) are allowed.

If administration of chemotherapy is delayed, there will be no dosemodification of GA101, and the administration of GA101 and all

chemotherapy drugs should be delayed for the same time frame, e.g., if miniCHOP therapy is delayed, administration of GA101 should also be delayed so that they are given on day 1 of the same cycles.

## Hematologic and Non-Hematologic Toxicities

Dosing of miniCHOP and GA101 may be resumed upon the resolution of <u>hematologic toxicity</u> to Grade  $\leq 2$  (platelets must resolve to Grade  $\leq 1$ ) or baseline status for the first episode.

For <u>non-hematologic toxicities</u>, dosing of GA101-miniCHOP-may only be resumed upon resolution to Grade ≤1 or baseline status.

For Grade  $\geq 2$  non-hematologic toxicities (excluding alopecia, nausea, and vomiting), treatment with GA101-miniCHOP will be delayed until resolution to Grade  $\leq 1$  (or baseline status for all except hemorrhagic cystitis), for a maximum of 21 days.

In addition, resumption of dosing without complete resolution of toxicity may only be considered after careful weighing of the risks and benefits with the patient and agreement between the investigator and the Sponsor.

If treatment is delayed for more than 21 days (except for hepatitis B reactivation), the patient will be withdrawn from study treatment (note that lymphopenia is not considered a cytopenic toxicity, as it is an expected outcome of therapy).

Patients who discontinue all study treatment for adverse events should remain on the study and continue to have disease assessments until progression and standard follow-up.

In the event of grade 2 neurological vincristine-related toxicity (sensory or motor polyneuritis, constipation, or visual or auditory changes) vincristine can be discontinued.

#### **Permitted concomitant therapies**

Prevention of tumour lysis syndrome by alkalinisation or hypouricaemic drugs is allowed if necessary.

Antiemetic therapy with SHT3 antagonists can be given at each cycle.



| | Patients will receive prophylactic treatment with Bactrim 2 cp/day twice a week during all the chemotherapy. CNS prophylaxis with intrathecal infusion of methotrexate and steroid is allowed according to local clinical practice (i.e. patients with testicular involvement or patients considered at high risk of CNS relapse). |
|---|---|
| | In patients HBcAb+, prophylaxis for hepatitis B reactivation with Lamivudine 100mg/die from the start of the treatment to one year after the end of the treatment is mandatory. |
| | Pre-medication for GA101 infusion with oral acetaminophen (e.g., 650–1000 mg) and an antihistamine such as diphenhydramine hydrochloride (50–100 mg) 30–60 minutes prior to starting each infusion (unless contraindicated). An additional glucocorticoid (e.g., 100 mg IV <i>prednisone or prednisolone</i> or equivalent) is allowed at the investigator's discretion. For patients who do not experience infusion-related symptoms with their previous infusion, pre-medication at subsequent infusions may be omitted at the investigator's discretion. |
| | Prophylaxis with levofloxacine or ciprofloxacine and fluconazole/itraconazole/posaconazole are allowed. Platelets and red blood cell transfusion are allowed, if needed. |
| Treatment duration | 6 months |
| Statistical methods: | The primary objective of the study is to demonstrate a clinical benefit in Complete Remission Rate (CRR) and safety with GA101-miniCHOP association in elderly unfit patients newly diagnosed with diffuse large B-cell lymphoma. For the purposes of this study, as the reference CR rate (Peyrade et al, Lancet Oncol – 2011) was defined with 1999 International Criteria for response (Cheson, JCO 1999), the response rate to therapy will be based on a Central Independent Review of response that will not consider the results of FDG-PET but will only use the conventional CT scan images. Response defined according to Cheson 2007 International Criteria will also be provided as study result. |
| The sample size has been estimated according to a optimal Simon design. The null hypothesis (p0) has been set equal <b>0.60</b> on the bas reported by F. Peyrade et al. With a type I (alfa) error of <b>0.10</b> (10%) and a type II (beta (power=90%) the alternative hypothesis (p1) is <b>0.75</b> , i.e. a CR rate the combination GA101-miniCHOP expected. A schema of the design is below reported. | |
| | R1 = 21 N1 = 34 R2 = 47 Ntot = 71 EN(p0) = 47 PET(p0) = 64.6% According to the two-stage design patients enrolment will proceed as follows: - the enrolment of 34 patients (stage 1) is planned: if at least 22 patients will achieve CR the study will continue; - additional 37 patients are entered (stage II): if at least 48 patients out of 71 will achieve a CR the study will be considered of possible evaluation for the efficacy of the treatment. |



| Considering a withdrawal rate of 10%, the enrollment may continue until <b>78</b> |
|---|
| patients are accrued in order to have at least 71 eligible patients. If GA101- |
| miniCHOP will be active, the probability to declare inactivity is 0.0964 and the |
| probability to stop the study at first stage is 0.0610. |

# **Study Flow Chart**

| Number | of | patients | 34 patients |
|----------|----|----------|-------------|
| planned | | | |
| Number | of | patients | 33 |
| analysed | | _ | |
| Number | of | excluded | 4 |
| patients | | | |



FIL\_GAEL\_FSR\_v.1.0\_April 30th, 2020

14 CR, 6 PR, 6 PD



# **Overall Study**

 Table 1: Overall Study and Treatment Administration

| | Therapy: GA101-miniCHOP |
|---|---|
| Started N. Patients enrolled 33 | |
| Completed | N. Patients that have completed therapy 26 |
| Not Completed | 7 |
| Lack of Efficacy | 19 |

**Table 2:** Demographic characteristic of enrolled patients (n=33)

| Variable | Median (2.5-97.5 percentile) |
|------------------------|------------------------------|
| Age, years | 82 (68-89) |
| Hb, g/dL | 12.9 (8.9-15.7) |
| WBC 10 <sup>9</sup> /l | 7.7 (3.6-20.5) |
| ALC 10 <sup>9</sup> /1 | 1.2 (0.2-3.5) |

| Variable | Status | N (%) |
|------------|--------|---------|
| Gender | M | 18 (55) |
| | F | 15 (45) |
| Stage | II | 6 (18) |
| | III | 11 (33) |
| | IV | 16 (48) |
| BM | - | 27 (82) |
| | + | 6 (18) |
| ECOG PS | 0 | 12 (35) |
| | 1 | 19 (58) |
| | 2 | 1 (3) |
| | 3 | 1 (3) |
| B-symptoms | Α | 27 (82) |
| | В | 6 (18) |
| Histology | DLBCL | 32 (97) |
| | T LBCL | 1 (3) |
| LDH | ≤ULN | 10 (30) |
| | >ULN | 23 (70) |
| B2M | ≤ULN | 2 (7) |
| | >ULN | 25 (93) |
| IPI | 0-1 | 4 (12) |
| | 2 | 8 (24) |
| | 3-5 | 21 (64) |
| CGA | UNFIT | 28 (85) |
| | FRAIL | 5 (15) |

Missing: ALC n=1, B2M n=6

DLBCL: diffuse large B-cell lymphoma, TLBCL: T-cell/histiocyte LBCL

WBC: white blood cell; ALC: absolute lymphocyte count; ULN: upper limit of normality; B2M: beta2-microglobuline; LDH lactate dehydrogenase; BM bone marrow involvement

interogradume, EDTI lactate deliyarogenase, Divi done marrow involv



# **Efficacy evaluation:**

Table 3. Complete remission (CR) rate according to Cheson 1999.

| | Final response | |
|----------|----------------|------------------|
| Response | N | % (95CI) |
| CR | 14 | 42.4 (25.5-60.8) |
| PR | 8 | 24.2 (11.1-42.3) |
| SD | 2 | 6.1 (0.7-20.2) |
| PD | 8 | 24.2 (11.1-42.3) |
| NA | 1 | 3.0 (0.1-15.8) |
| Total | 33 | |

CR: complete remission, PR: partial remission, SD: stable disease, PD: progression disease, NA: not assessed.

95CI: 95% confidence interval (Clopper-Pearson)

NA: one patents withdrawal after 1 cycle due fever hospitalization.

# # CR 14: it does not exceed the threshold of 21 CR as expected from the optimal Simon two stage. Interim analysis failed for efficacy.

Table 4. Dose Intensity (mean, 95%CI) according to Hryniuk.

| Cycles | GA101 | Doxorubicin | Cyclophosphamide | Vincristine |
|---|---|---|---|---|
| 1-4 | 0.94 (0.92-0.96) | 0.93 (0.90-0.95) | 0.93 (0.90-0.95) | 0.94 (0.91-0.96) |
| 5-8 (6) | 0.99 (0.95-1.04) | 0.98 (0.95-1.01) | 0.97 (0.94-1.00) | 0.98 (0.93-1.03) |

# **Safety Evaluation:**

**Table 5.** Hematological and extra-hematological adverse events (AE). Maximum adverse event collected during induction treatment (n=33).



| Adverse Event - Haematological | Grade 1-2 | | Grad | Grade 3-4 |
|---|---|---|---|---|
| | n | % | n | % |
| Anemia | 6 | 18,2 | 0 | 0,0 |
| Leukopenia | 2 | 6,1 | 2 | 6,1 |
| Neutropenia | 2 | 6,1 | 13 | 39,4 |
| Piastrinopenia | 10 | 30,3 | 1 | 3,0 |
| Febrile neutropenia | 0 | 0,0 | 0 | 0,0 |
| Adverse Event - Non-heamatological | Grad | Grade 1-2 Grade 3- | | le 3-4 |
| | n | % | n | % |
| Cardiac disorders | 3 | 9,1 | 2 | 6,1 |
| Congenital/familial/genetic disorders | 0 | 0,0 | 0 | 0,0 |
| Ear and labyrinth disorders | 0 | 0,0 | 0 | 0,0 |
| Endocrine disorders | 0 | 0,0 | 0 | 0,0 |
| Eye disorders | 0 | 0,0 | 0 | 0,0 |
| Gastrointestinal disorders | 11 | 33,3 | 1 | 3,0 |
| General disorders and administration site conditions | 4 | 12,1 | 2 | 6,1 |
| Hepatobiliary disorders | 0 | 0,0 | 2 | 6,1 |
| Immune system disorders | 0 | 0,0 | 0 | 0,0 |
| Infections | 6 | 18,2 | 1 | 3,0 |
| Injury/poisoning/procedural complications | 0 | 0,0 | 2 | 6,1 |
| Investigations | 2 | 6,1 | 1 | 3,0 |
| Metabolism and nutrition disorders | 5 | 15,2 | 3 | 9,1 |
| Musculoskeletal and connective tissue disorders | 5 | 15,2 | 3 | 9,1 |
| Neoplasms benign/malignant/unspecified | 0 | 0,0 | 2 | 6,1 |
| Nervous system disorders/Psychiatric disorders | 6 | 18,2 | 1 | 3,0 |
| Pregnancy/puerperium and perinatal conditions | 0 | 0,0 | 0 | 0,0 |
| Renal and urinary disorders | 2 | 6,1 | 0 | 0,0 |
| Reproductive system and breast disorders | 0 | 0,0 | 0 | 0,0 |
| Respiratory/thoracic and mediastinal disorders | 5 | 15,2 | 0 | 0,0 |
| Skin and subcutaneous tissue disorders | 0 | 0,0 | 0 | 0,0 |
| Social circumstances | 0 | 0,0 | 0 | 0,0 |
| Surgical and medical procedures | 0 | 0,0 | 0 | 0,0 |
| Vascular disorders | 1 | 3,0 | 0 | 0,0 |
| Other (specify) | 8 | 24,2 | 0 | 0,0 |

One patient was dead after with heart failure grade 4



| Collected ad Other toxicities (n=8) - | |
|---------------------------------------|---|
| description | |
| Epigastric pain | 2 |
| Dysgeusia | 1 |
| Fever | 2 |
| Infusion reaction | 2 |
| Asthenia; bone pain | 2 |
| Infiammatory edema | 1 |
| Fever | 2 |
| Pain | 2 |

**Table 6.** List of serious advent events (SAE)

| ID | Date of Onset SAE/SUSAR | Report (I or FU | Event Short Description | Gravity of the event | Outcome of the event at report time | Relationship | Suspected Drug |
|---|---|---|---|---|---|---|---|
| 0002GAEL | 20/12/2015 SAE | | nausea | Caused/Prolonged Hospitalisation | Not Recovered/Not Resolved | Unrelated | none |
| 0002GAEL | 19/02/2016 SAE | 1 | femure fracture | Caused/Prolonged Hospitalisation | Not Recovered/Not Resolved | Unrelated | none |
| 0002GAEL | 19/02/2016 SAE | FU | femure fracture | Caused/Prolonged Hospitalisation | Recovered/Resolved | Unrelated | none |
| 0002GAEL | 31/03/2016 SUSAR | ı | congestive heart failure | Caused/Prolonged Hospitalisation | Not Recovered/Not Resolved | Unrelated | none |
| 0002GAEL | 22/06/2016 SAE | I/FU | congestive heart failure | Death | Fatal | Possible | GA101 |
| 0004GAEL | 08/12/2015 SAE | ı | lumbar pain, vertebral collapse | Caused/Prolonged Hospitalisation | Not Recovered/Not Resolved | Unrelated | obinutuzumab miniCHOP |
| 0005GAEL | 08/02/2016 SAE | ı | fever | Caused/Prolonged Hospitalisation | Not Recovered/Not Resolved | Unrelated | obinutuzumab miniCHOP |
| 0005GAEL | 08/02/2016 SAE | FU | sepsis | Caused/Prolonged Hospitalisation | Recovered/Resolved | Unrelated | none |
| 0005GAEL | 07/08/2016 SAE | I/FU | sepsis | Death | Fatal | Unrelated | |
| 0015GAEL | 15/04/2016 SAE | | BPCO - Heart Failure | Caused/Prolonged Hospitalisation | Not Recovered/Not Resolved | Probable | obinutuzumab miniCHOP |
| 0026GAEL | 09/05/2017 SUSAR | _ | breast cancer | Other medically important condition | Not Recovered/Not Resolved | Unrelated | GA101 |
| 0026GAEL | 09/05/2017 SUSAR | FU | breast cancer | Other medically important condition | Not Recovered/Not Resolved | Unrelated | doxorubicina, vincristina, ciclofosfamide |
| 0026GAEL | 09/05/2017 SUSAR | FU | breast cancer | Other medically important condition | Not Recovered/Not Resolved | Unrelated | prednisone |
| 0026GAEL | 19/07/2017 SUSAR | l | non small cell lung cancer | Other medically important condition | Unknown | Unrelated | obinutuzumab |
| 0026GAEL | 19/07/2017 SUSAR | FU | non small cell lung cancer | Other medically important condition | Unknown | Unrelated | obinutuzumab/vincristina/doxorubicina/ciclofosfamide |
| 0026GAEL | 19/07/2017 SUSAR | FU | non small cell lung cancer | Other medically important condition | Unknown | Unrelated | prednisone |
| 0032GAEL | 16/06/2016 SAE | ı | Fever | Caused/Prolonged Hospitalisation | Not Recovered/Not Resolved | Possible | GA101 |
| 0036GAEL | 16/06/2016 SAE | ı | Atrial fibrillation | Caused/Prolonged Hospitalisation | Unknown | Unrelated | not started |
| 0036GAEL | 18/06/2016 SAE | FU | Atrial fibrillation - sepsi due to Klebsiella Pneumoniae | Caused/Prolonged Hospitalisation | Fatal | Possible | not started |

I: Initial; FU: adverse event follow-up

ID 0036: SAE recorded before starting 1st cycle of treatment. Not included in the 33 evaluable patients.

ID 0026: SUSAR during follow-up post induction.

SAE/SUSAR reported in 7 patients (Six evaluated and one exit before treatment).

## **Secondary End-Point**

**Overall Response Rate (ORR: CR+PR):** 67% (95%CI 48-82%)

**Overall survival (OS):** After a median of 32 months (95%CI 15-38 months), from the date of registration in the study, were observed 11 death: 7 for progression of disease, 1 for probable progression of lymphoma, 1 for heart failure, 1 for sepsis and one due unknown cause.

The 24-months OS% was 69% (95%CI 50-82%).

Progression Free Survival (PFS): Were observed 17 events, with a 24-months PFS of 53% (34-68%).





## **Summary – Conclusions:**

In conclusion, our phase II study confirmed the activity and safety of Ga101-miniCHOP for the treatment of older, unfit patients with DLBCL, but was not able to show it as a promising regimen to challenge the current standard R-miniCHOP. To improve treatment efficacy in this hard to-treat patient population, different strategies should be adopted that include better patient and/or lymphoma profiling and the use of new drugs with a novel non-cross-resistant mechanism of action.

We attest the accuracy and truthfulness of the information contained in this Report.

Date of report: April 30th, 2020

Dr. Francesco Merli

Principal Investigator and

President of Fondazione Italiana Linfomi